CLINICAL TRIAL: NCT02456337
Title: Xenogenous Collagen Matrix Graft Associated or Not With Enamel Matrix Derivative Proteins in the Treatment of Gingival Recession Class I and II of Miller: Randomized Controlled Clinical Study
Brief Title: Xenogenous Collagen Matrix Graft With or Without Enamel Matrix Proteins Derivative for Root Coverage
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Campinas, Brazil (Other)
Collaborators: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Enilson Antonio Sallum, Professor. Department of Periodontics. Piracicaba Dental School. State University of Campinas (UNICAMP), Piracicaba, São Paulo, Brazil., University of Campinas, Brazil
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 067/2013; 2013/19473-6 (Other Grant/Funding Number: FAPESP)
Record Dates: First submitted 2015-05-25; First posted 2015-05-28 (Estimated); Last update posted 2016-10-27 (Estimated); Status verified 2015-12

CONDITIONS: Gingival Recession
Keywords: Gingival Recession; Coronally advanced flap; Periodontal regeneration
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- CAF+MC+EMD (Experimental): Coronally Advanced Flap with Mucograft and Emdogain
  Interventions: Device: Mucograft; Device: Emdogain; Procedure: Coronally Advanced flap
- CAF+MC (Active Comparator): Coronally Advanced Flap with Mucograft
  Interventions: Device: Mucograft; Procedure: Coronally Advanced flap
- CAF+EMD (Active Comparator): Coronally Advanced Flap with Emdogain
  Interventions: Device: Emdogain; Procedure: Coronally Advanced flap
- CAF (Active Comparator): Coronally Advanced Flap alone
  Interventions: Procedure: Coronally Advanced flap

INTERVENTIONS:
Device: Mucograft — Coronally advanced flap associated to Xenogenous collagen matrix graft (mucograft) for the treatment of gingival recessions Miller Class I or II.
  Arms: CAF+MC; CAF+MC+EMD
Device: Emdogain — Coronally advanced flap associated to Enamel Matrix Derivative (Emdogain) for the treatment of gingival recessions Miller Class I or II.
  Arms: CAF+EMD; CAF+MC+EMD
Procedure: Coronally Advanced flap — Coronally advanced flap for the treatment of gingival recessions Miller Class I or II.

SUMMARY:
The purpose of this study is to evaluate the reduction of gingival recession of single Miller Class I and II defects treated by coronally advanced flap with subepithelial porcine collagen matrix graft and / or enamel matrix proteins.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Presence of at least one Class I or II Miller gingival recession ≥ 2.5 mm in maxillary canines or premolars with identifiable cementum-enamel junction (CEJ) and without deep non-carious cervical lesions (< 0.5 mm): A +(Pini-Prato et al. 2010).
* Aesthetic complaint and/or presence of dentin hypersensitivity to air stimulus.
* Full-mouth visible plaque index ≤ 20% (Ainamo & Bay 1975).
* Full-mouth sulcus bleeding index ≤ 20% (Mühlemann & Son 1971).

Exclusion Criteria:

* Smoking.
* Pregnancy.
* Presence of systemic disorders (diabetes, hypertension, heart disease or any other condition that could contraindicate periodontal surgery).
* Use of medications (immunosuppressants, phenytoin or anything else that might affect mucosal healing and repair).
* Previous periodontal surgery in the area.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 49 (Actual)
Dates: Start 2014-07; Primary Completion 2016-09 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Recession Reduction | 6 months
  Measured as a difference between gingival margin between gingival recession depth at baseline and gingival recession at 6 months follow-up.

SECONDARY OUTCOMES:
Complete root coverage | 6 months
  Assessed as percentage of sites with complete root coverage

OTHER OUTCOMES:
Keratinized tissue thickness | 6 months
  Measured at a midpoint between gingival margin and mucogingival junction using a endodontic spreader pierced perpendicular and through the soft tissue

CONTACTS AND LOCATIONS:
Overall Officials: Enilson A Sallum, PhD, Study Chair — University of Campinas
Locations (1):
- Piracicaba Dental School, State University of Campinas, Piracicaba, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sangiorgio JPM, Neves FLDS, Rocha Dos Santos M, Franca-Grohmann IL, Casarin RCV, Casati MZ, Santamaria MP, Sallum EA. Xenogenous Collagen Matrix and/or Enamel Matrix Derivative for Treatment of Localized Gingival Recessions: A Randomized Clinical Trial. Part I: Clinical Outcomes. J Periodontol. 2017 Dec;88(12):1309-1318. doi: 10.1902/jop.2017.170126. Epub 2017 Jul 28. PMID 28753100